CLINICAL TRIAL: NCT00000189
Title: Gepirone vs Placebo in Treatment of Cocaine Dependence
Brief Title: Gepirone vs Placebo in Treatment of Cocaine Dependence - 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, James Cornish, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-00144-3; 3R01DA012268 (NIH); K20-00144-3
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine Dependence; Gepirone
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — gepirone

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Gepirone

SUMMARY:
The purpose of this study is to test antidepressant medication, gepirone, as a pharmacotherapy for cocaine dependent subjects.

ELIGIBILITY:
Please contact site for information.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 1990-01; Primary Completion 1991-02 (Actual); Study Completion 1991-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Cornish, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Jenkins SW, Warfield NA, Blaine JD, Cornish J, Ling W, Rosen MI, Urschel H 3rd, Wesson D, Ziedonis D. A pilot trial of gepirone vs. placebo in the treatment of cocaine dependency. Psychopharmacol Bull. 1992;28(1):21-6. PMID 1609038